CLINICAL TRIAL: NCT04760522
Title: Genome-based Management of Patients in Precision Medicine (Ge-Med) Towards a Genomic Health Program
Acronym: GE-MED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GE-MED APPROACH
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Rare Diseases; Genetic Predisposition to Disease
Keywords: Rare Diseases; Genetic Predisposition; Whole Exome Sequencing (WES); Whole Genome Sequencing (WGS); Familial cancer syndromes; Polygenic Risk Scores (PRS)
MeSH Terms: conditions — Rare Diseases; Genetic Predisposition to Disease; Genetic Risk Score

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WGS Diagnostic (Experimental): Both underage and adult persons (male and female) with diagnostically unsolved rare diseases who have been or are included into diagnostic care at the University Hospital Tübingen, Germany (UKT) and who are suspected of having a genetic cause of the disease.
  Study related procedures: Blood sampling, anamnesis including pedigree, Next Generation Sequencing (NGS) analysis and other omics analysis (transcriptomics, proteomics, metabolomics).
  Interventions: Genetic: WGS Diagnostic: Blood take for genetic diagnostic

INTERVENTIONS:
Genetic: WGS Diagnostic: Blood take for genetic diagnostic — Blood sampling, short clinical characterization, WGS based sequencing, NGS analysis and other omics analysis (transcriptomics, proteomics, metabolomics).

SUMMARY:
The GE-MED APPROACH project will enroll patients (n = appr. 12.000) with unclear molecular cause of the disease, suspected genetic cause of the disease without detailed molecular analysis like Whole Exome Sequencing (WES).

The novelty of this study is to integrate genomic health concepts into immediate clinical care. To achieve these goals, a novel structure for the Triple P (3P) concept of personalized medicine (Personalized, Predictive, Preventive) integrated into a well-established health care system and associated with novel decentralized Disease Analysing Task Forces (DATF) will be implemented.

The overall goal of this study is to implement, for the first time, Whole Genome Sequencing (WGS) analysis as a first line diagnostic test for all clinical indications such as Rare Disease (RD )and familial cancer syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Unclear molecular cause of the disease
* Suspected genetic cause of the disease

Exclusion Criteria:

* Missing informed consent of the patient and if applicable the legal representative
* Previously performed WES or panel analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of WGS analysis | Day 1
  WGS analysis as a first line diagnostic test for all clinical indications

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Rieß, Prof. Dr., Study Director — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The GE-MED APPROACH study will provide data in a pseudonymized manner to national and international databases set up to increase the diagnostic yield through advanced analysis tools and matchmaking against other cohorts
Supporting Information: Analytic Code
Time Frame: Data will become available after analysis and unlimited.
Access Criteria: Authorized users within the participating organizations.